CLINICAL TRIAL: NCT04564235
Title: Risk of Recurrence of de Novo Mutations: Research and Quantification of Paternal Germinal Mosaicism by the Combined Use of Genomic Tools
Acronym: RRMUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/0401/HP
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Developmental Disorders
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indication for a genome-wide analysis in the proband (Experimental)
  Interventions: Genetic: genome-wide analyses; Genetic: Search for de novo mutations in paternal sperm samples

INTERVENTIONS:
Genetic: genome-wide analyses — genome-wide analyses will be done in patients and parents (father, mother)
Genetic: Search for de novo mutations in paternal sperm samples — Sperm analysis will be done in paternal samples

SUMMARY:
1. Inclusion of 5 families Inclusions will be made by the clinical genetics department of the Rouen University Hospital (monocentric study) and will correspond to trios of parents + child with unexplained developmental abnormalities. The inclusion of patients will be integrated in routine care and will have as immediate benefit for the included families the extensive analysis of the proband and their parents' genomes by short and long read sequencing techniques, which represent the most comprehensive diagnostic tests for developmental diseases, and which are not currently routinely available. Inclusion in clinical genetics by clinicians accustomed to prescribing genome-wide analyses will allow clear and complete information to families. Collection of consents. The trio's DNA will already be available at the molecular genetics laboratory, and a new blood sample may be proposed if necessary. Collection of sperm from the father.
2. Identification of a large set of de novo mutations. Extraction of blood DNA and sending for sequencing of the complete genome to the National Centre for Research in Human Genomics (CNRGH, Evry), in the framework of a collaboration already initiated. Analysis of the sequencing data thanks to the already existing expertise in Rouen. Identification of about 40-120 de novo mutations per trio. At this stage: interpretation of the variations identified with the secondary objective of identifying the cause of the disease in children. Long read genomes will allow to phase the de novo variants to the paternal or to the maternal haplotype.
3. Search for de novo mutations in paternal sperm samples. Extraction of spermatic DNA. Design of a sequencing panel targeting the genetic variations identified in the different trios. Preparation of the libraries, targeted high throughput sequencing at great depth thanks to the techniques and equipment already operational. Specific search for the de novo variations identified in the probands (in 2.), with for each evaluation of (i) the presence of the variation in the sperm sample, (ii) the quantity of mosaicism, reflecting the proportion of carrier spermatozoa and therefore the risk of recurrence, (iii) the presence of my variation in the blood sample of both parents in deep sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Trio consisting of a child with a developmental disorder and both unaffected parents
* Absence of etiology after clinical expertise and genetic testing
* Indication of a genome-wide sequencing analysis
* Child from spontaneous pregnancy without ovulation stimulation treatment
* Availability of DNA blood samples
* Affiliation to a social insurance
* Patient or patient's legal representative who has read and understood the information letter and has signed the consent form

Exclusion Criteria:

* Lack of indication for a genome-wide analysis in the proband
* Etiology of the developmental disorder already identified
* Proband born after In-Vitro Fertilization
* Impossibility of non-invasive sperm collection from the father

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Proportion of the patient's de novo mutations detectable in the father's sperm | Day 1

SECONDARY OUTCOMES:
Number of patients for whom molecular diagnosis has been obtained (cause of developmental disability identified) ≥1 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: François LECOQUIERRE, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No